CLINICAL TRIAL: NCT06259474
Title: Effect of Intraabdominal Hypopressive Exercises on Postnatal Backache and Functional Disability
Brief Title: Effect of Hypopressive Exercises on Postpartum Backache and Functional Disability
Acronym: LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Salwa A. Shawat, Principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hypopressive Exerrcises
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: Hypopressive Exercises
MeSH Terms: conditions — Low Back Pain | interventions — Diathermy; Dosage Forms

STUDY DESIGN:
Intervention Model Description: The study was designed as randomized, single blind pretest and posttest controlled trial. Approval was granted by the Ethical Committee of the Faculty of Physiotherapy at Kafr El Sheikh University under the number (T/ WH /2/2023/38). Each participant signed a written informed consent agreeing to adhere to the treatment plan for two months after discussing the benefits, goals and strategy of this study. They were also free to leave the study whenever they wished, for any reason. The principal investigator placed copies of the subjects' numbers in a vase and randomly assigned them to groups (A, B).
  2.2. Subjects
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group (A): 20 subjects combined HE with traditional treatments for low back pain (heat therapy, medication, and progressive strength training).
  Interventions: Combination Product: Hypopressive Exercises and (heat therapy, medication, and progressive strength training)
- Group B (Active Comparator): Group (B) :20 subjects received the same conventional treatment for low back pain as group (A), including heat therapy, medication, and progressive strength training.
  Interventions: Combination Product: Hypopressive Exercises and (heat therapy, medication, and progressive strength training)

INTERVENTIONS:
Combination Product: Hypopressive Exercises and (heat therapy, medication, and progressive strength training) — 20 subjects combined HE with traditional treatments for LBP (heat therapy, medication, and progressive strength training). Each session consisted of 5 to 10 HEs. Participants were instructed not to hold their breath or perform PFMS contractions during the HEs. Traditional treatment for low back pain typically involved using medications like acetaminophen (0.5-1 g three times daily) and heat therapy, which consisted of using a continuous heat wrap for 2 hours, 3 times per week at 40 °C, one hour before and after the session
  Other Names: Hypopressive abdominal gymnastics

SUMMARY:
The purpose of this study was to evaluate the effectiveness of hypopressive exercise in postpartum females with abnormal hyperlordosis and back pain.

DETAILED DESCRIPTION:
More than half of new mothers suffer from lower back pain , with one-third of these occurring within three months of delivery. In addition, 40% of women report moderate to severe disability due to this pain . Persistent low back pain not only causes discomfort, but can also lead to a lower quality of life, decreased fitness levels, and fear of exercise. Women with chronic low back pain may find it difficult to manage housework, hobbies, and work . Stress, both physical and psychological, triggers the release of cortisol by the hypothalamic-pituitary-adrenal axis (HPAA) to suppress inflammation. If left untreated, low back pain can cause cortisol dysfunction, inflammation, and pain . Excessive pain can interfere with milk transfer in lactating women, while medical trreatments as sedating medications can cause respiratory depression in infants . Studies have shown that age, gender, pregnancy, and obesity may influence the degree of lumbar lordosis which can lead to postural pain, radiculopathy, and facet joint pain . Changes in the curvature and spinal segments of the anterior-posterior axis contribute to the unloading of the pelvic organs by sympathetic (T10-L2) and parasympathetic (S2-S4) nerves, resulting in a lower pain threshold. The birthing process exerts the most pressure on the hip joint, pelvis, and abdominal muscles, which in turn affects the back, pelvis, and sacroiliac joints. Vaginal birth has been found to affect the strength and stiffness of the pelvic floor . The still enlarged levator hiatus is unable to withstand the increased pressure on the abdomen, which may lead to the development of several disorders in the future . Physical therapy, stabilization belts, nerve stimulation, medications, acupuncture, massage, relaxation techniques, and yoga are all viable options for treating low back pain. Weight loss has been shown to decrease the likelihood and severity of low back pain (Bailey, 2009). While conventional treatments such as medications or surgery, while promising, are also associated with significant side effects, such as diarrhea, nausea, vomiting, leg cramps or other muscle spasms, insomnia, headaches, and abnormal dreams.

The American College of Obstetricians and Gynecologists (ACOG) points out that exercise is a good way to reduce stress, prevent postpartum depression, increase energy, strengthen and tone abdominal muscles, and promote better sleep . The diaphragm and pelvic floor are synergistic muscles that work with the transversus abdominis to maintain intra-abdominal pressure and maintain various postures .

Theoretically, the goal of HE is to decrease intra-abdominal pressure, while the basal tone of the deep abdominal muscles and pelvic floor muscles (PFM) is increased without conscious activation . The authors claim that a decrease in abdominal pressure with a latency of a few seconds triggers type I reflex activity in the abdominal wall and pelvic floor muscles. These exercises gradually activate the abdominal and pelvic floor muscles and cause direct activation of the transversus abdominal muscle, which strengthens the abdominal girdle, stabilizes the spine , and contracts bilaterally, forming fascial bands that contract like a brace . This deep muscle contributes to stability in three ways: it modulates intra-abdominal pressure, transmits force to the lumbar spine via the thoracolumbar fascia, and increases lumbar spine stiffness Considering the current stage of maternal life, we aimed to determine the effects of this exercise on low back pain, functional limitations, and lumbar angle.

ELIGIBILITY:
Inclusion Criteria:

Participants must have a healthy pregnancy Normal vaginal birth LBP that existed 24 weeks after giving birth Functional limitations in daily activities. Participants' age from 20 to 35 years

Exclusion Criteria:

* No more than two prior pregnancies BMI of less than 25 kg/m2 to participate. Women who were under pharmacological or psychological treatment, had pelvic tumors, lumbar disk herniation, heart disease, hypertension, lumbar spine tumors, chronic uterine prolapse, chronic pelvic pain, lumbar spondylosis, or lumbar spondylolisthesis.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain | Once at the start and once at the end of the stufy
  The Revised Short McGill Pain Questionnaire consists of 22 pain descriptions rated on a scale from 0 to 10. A score of 0 indicates no pain, whereas a score of 10 represents the most severe pain ever experienced by the patient. The questionnaire includes four subscales. The four subacales were combined to create an overall score, with higher scores indicating greater discomfort.

SECONDARY OUTCOMES:
Assessment of functional disability | Once at the start and once at the end if the study
  The Patient-Specific Functional Scale (PSFS) assessed functional changes in patients with musculoskeletal illnesses using self-reported data. Patients rated to five activities on an 11-point scale based on their current level of difficulty.The Patient-Specific Functional Scale (PSFS) assessed functional changes in patients with musculoskeletal illnesses using self-reported data. Patients rated to five activities on an 11-point scale based on their current level of difficulty
Assessment of lumbar lordotic angle | Once at the start and once at the end if the study
  The angle was measured using flexible ruler once before and once after the study by the primary examiner, who repeated each measurement three times.The angle was determined by calculating the lengths of the h and L lines and using the formula θ=4 arc tan 2 h/L

IPD SHARING:
Plan to Share IPD: Undecided